CLINICAL TRIAL: NCT04616820
Title: Venous Pulmonary Compared to Venous Systemic Blood Level of Endocan During On-pump Cardiac Surgery
Brief Title: Endocan Blood Level in Pulmonary Circulation
Acronym: ENDOPULM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Biothelis (Unknown)
Responsible Party: Sponsor
Other Study IDs: ENDOPULM
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; Lung
Keywords: Endocan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endocan blood levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endocan is a proteoglycan produced by the vascular endothelium. Animal studies suggested that the synthesis mainly happen in the pulmonary circulation, but this hypothesis has never been confirmed in humans.

DETAILED DESCRIPTION:
The investigators will measure endocan levels in both pulmonary and systemic venous blood in patients undergoing on pump cardiac surgery.

The main objective is to quantify the difference of endocan blood level between the pulmonary and the systemic circulation.

ELIGIBILITY:
Inclusion Criteria:

* Planned on pump coronary artery bypass surgery
* Non opposition

Exclusion Criteria:

* Age < 18 years old
* Emergent surgery
* Valvular replacement surgery
* Combined cardiac surgery
* Patients with inflammatory, infectious or evolutive neoplastic pulmonary disease
* Patients with valvular problems, in particular aortic insufficiency
* Patients who refuse to participate
* Legal inability or disability
* Patients who will probably not cooperate for the study
* Pregnancy and/or breast feeding
* Patients not in the Social security system
* Patients in the exclusion period of another study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients who are sheduled for on-pump coronary artery bypass surgery in the Cardiac Surgery Department of the University Hospital of Besancon.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Quantify the difference of Endocan blood levels between pulmonary and systemic circulation at the end of cardiopulmonary bypass | At the end of cardiopulmonary bypass
  Blood samples will be collected at the same time in both pulmonary and systemic circulation at the end of cardiopulmonary bypass to measure Endocan blood level. The primary outcome will be the absolute difference between the Endocan blod level in the pulmonary circulation and in the systemic circulation.

SECONDARY OUTCOMES:
Kinetic of Endocan blood level in the systemic circulation during on pump cardiac surgery | Prior to the start of cardiopulmonary bypass, at the beginning and at the end of cardiopulmonary bypass, and at the end of surgery
  Blood samples will be collected in the systemic circulation prior to the start of cardiopulmonary bypass, at the beginning of the cardiopulmonary bypass and at the end of cardiopulmonary bypass, and at the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEBAT, Study Chair — CHU Jean Minjoz Besançon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lassalle P, Molet S, Janin A, Heyden JV, Tavernier J, Fiers W, Devos R, Tonnel AB. ESM-1 is a novel human endothelial cell-specific molecule expressed in lung and regulated by cytokines. J Biol Chem. 1996 Aug 23;271(34):20458-64. doi: 10.1074/jbc.271.34.20458. PMID 8702785
- [Background] Kao SJ, Chuang CY, Tang CH, Lin CH, Bien MY, Yu MC, Bai KJ, Yang SF, Chien MH. Plasma endothelial cell-specific molecule-1 (ESM-1) in management of community-acquired pneumonia. Clin Chem Lab Med. 2014 Mar;52(3):445-51. doi: 10.1515/cclm-2013-0638. PMID 24108208
- [Background] Palud A, Parmentier-Decrucq E, Pastre J, De Freitas Caires N, Lassalle P, Mathieu D. Evaluation of endothelial biomarkers as predictors of organ failures in septic shock patients. Cytokine. 2015 Jun;73(2):213-8. doi: 10.1016/j.cyto.2015.02.013. Epub 2015 Mar 17. PMID 25794660
- [Background] Mikkelsen ME, Shah CV, Scherpereel A, Lanken PN, Lassalle P, Bellamy SL, Localio AR, Albelda SM, Meyer NJ, Christie JD. Lower serum endocan levels are associated with the development of acute lung injury after major trauma. J Crit Care. 2012 Oct;27(5):522.e11-7. doi: 10.1016/j.jcrc.2011.07.077. Epub 2011 Sep 29. PMID 21958978
- [Background] Mangat M, Amalakuhan B, Habib S, Reyes LF, Hinojosa CA, Rodriguez AH, Soni NJ, Anzueto A, Levine SM, Peters JI, Aliberti S, Sibila O, Rello J, Witzenrath M, Waterer GW, Martin-Loeches I, Blanquer J, Sanz F, Marcos PJ, Sole-Violan J, Chalmers JD, Feldman C, Wunderink RG, Cruz CSD, Orihuela CJ, Restrepo MI. High endocan levels are associated with the need for mechanical ventilation among patients with severe sepsis. Eur Respir J. 2017 Jul 5;50(1):1700013. doi: 10.1183/13993003.00013-2017. Print 2017 Jul. No abstract available. PMID 28679609
- [Background] Poinsot PA, Barrucand B, Ecarnot F, Lassalle P, Besch G, Chocron S, Perrotti A. Kinetics of endocan in patients undergoing cardiac surgery with and without cardiopulmonary bypass. Cytokine. 2018 Oct;110:328-332. doi: 10.1016/j.cyto.2018.03.040. Epub 2018 Apr 4. PMID 29627158
- [Background] Perrotti A, Chenevier-Gobeaux C, Ecarnot F, Bardonnet K, Barrucand B, Flicoteaux G, Lassalle P, Chocron S. Is Endocan a Diagnostic Marker for Pneumonia After Cardiac Surgery? The ENDOLUNG Study. Ann Thorac Surg. 2018 Feb;105(2):535-541. doi: 10.1016/j.athoracsur.2017.07.031. Epub 2017 Nov 11. PMID 29132699
- [Background] Madhivathanan PR, Fletcher N, Gaze D, Thomson R, Chandrasekaran V, Al-Subaie N, Valencia O, Sharma V. Perioperative kinetics of endocan in patients undergoing cardiac surgery with and without cardiopulmonary bypass. Cytokine. 2016 Jul;83:8-12. doi: 10.1016/j.cyto.2016.03.006. Epub 2016 Mar 19. PMID 26999704